CLINICAL TRIAL: NCT05871606
Title: Inhaled Nitric Oxide in Acute Ischemic Stroke Patients Undergoing Mechanical Thrombectomy: A Phase I Drug Pilot Research Plan
Brief Title: Inhaled Nitric Oxide in Acute Ischemic Stroke Patients Undergoing Mechanical Thrombectomy
Acronym: iNO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00090271
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Cerebrovascular Disorders; Acute Cerebrovascular Disease
Keywords: Stroke; blood clot extraction; large vessel occlusion
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Intervention Model Description: The study has been designed to follow a standard 3+3 cohort expansion design, assessing 5 doses. Specifically, 3 individuals will begin at dose 1. If none of these individuals experience a dose limiting toxicity (DLT), then the dose will be escalated to dose 2. DLT is defined as a patient experiencing sICH, our primary outcome measure, or any other listed ASE. Dose escalation will continue after each set of 3 individuals until at least one person experiences DLT. If only 1 of the 3 experience a DLT, the cohort will be expanded to 6 (an additional 3). If 2 of the 6 experience DLTs, then dose escalation is stopped and the previous dose level (one level below) is declared the maximum tolerated dose. If 2 of the initial 3 experience DLT, the previous dose level (one level below) is declared the maximum tolerated dose. However, if only 1 of 6 experience DLT, the dose will escalate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose 2 Group (Experimental): Dose 2- Inhaled Nitrous Oxide (iNO) 40ppm.
  Interventions: Drug: iNO
- Dose 3 Group (Experimental): Dose 3- Inhaled Nitrous Oxide (iNO) 50ppm.
  Interventions: Drug: iNO
- Dose 4 Group (Experimental): Dose 4- Inhaled Nitrous Oxide (iNO) 60ppm.
  Interventions: Drug: iNO
- Dose 5 Group (Experimental): Dose 5- Inhaled Nitrous Oxide (iNO) 70ppm.
  Interventions: Drug: iNO
- Dose 6 Group (Experimental): Dose 6- Inhaled Nitrous Oxide (iNO) 80ppm.
  Interventions: Drug: iNO
- Dose 1 Group (Experimental): Dose 1- Inhaled Nitrous Oxide (iNO) 20ppm.
  Interventions: Drug: iNO

INTERVENTIONS:
Drug: iNO — Inhaled Nitrous Oxide
  Other Names: Inhaled Nitrous Oxide

SUMMARY:
The purpose of this study is to determine the safety and feasibility of using inhaled nitric oxide (iNO) in patients undergoing intra-arterial mechanical thrombectomy (blood clot extraction or IAMT) for treatment of acute ischemic (non-bleeding) stroke (AIS).

DETAILED DESCRIPTION:
This dose escalation phase I study is to evaluate the safety and feasibility of iNO as adjunctive therapy in the treatment of AIS in adult patients with clinically significant strokes.

iNO will act as a selective vasodilator to ischemic tissues in the brain, increasing perfusion to the area of the brain most at risk (penumbra) in AIS patients. This therapy will help to increase collateral circulation and perfusion to the penumbra, salvaging this tissue and limiting the volume of core infarct while mitigating reperfusion injury to the salvaged tissue.

Protection of ischemic penumbra is paramount in IAMT stroke patients. IAMT to re-establish blood flow during AIS from a large vessel occlusion (LVO) reduces death and disability. Initially this intervention was recommended up until 6 hours after symptom onset, but more recently has proven safe and effective up to 16 and 24 hours after stroke onset in select patients. These studies have confirmed the long believed thought that supporting ischemic penumbra during AIS helps limit the size of the ultimate core infarct and therefore reduces disability and death from stroke. Treatment aimed at protecting ischemic penumbra is thus paramount to treatment and research endeavors in AIS patients.

iNO protects ischemic penumbra. Nitric oxide is an endothelial-derived vasodilator and has been shown to mediate cytoprotection after ischemic reperfusion injury and appears to aid in ischemic preconditioning signaling pathways. iNO has been shown to cause selective dilation of arterioles in the ischemic penumbra of stroke and subarachnoid hemorrhage animal models, helping augment the cerebral microcirculation and improve penumbral blood flow. This has been shown to reduce ischemic brain damage, limit core infarct, and consistently improve neurological outcome in a middle cerebral artery AIS mouse model

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and < 80
* Clinical evidence of acute ischemic (non-bleeding) stroke (AIS) with NIH Stroke Scale of 6 or higher
* Non-contrast Computed tomography (CT) Head with ASPECT (Alberta Stroke Program Early CT) score 6
* Symptom onset began < 16 hours from initiation of intra-arterial mechanical thrombectomy (IAMT) procedure
* CT Angiogram (CTA) evidence of anterior circulation MCA (Middle Cerebral Artery) M1 segment occlusion.
* CT Perfusion (CTP) evidence of core infarct volume of < 70ml and a ratio of ischemic tissue to initial core infarct volume of 1.8 or greater, and an absolute volume of penumbra of 15ml or greater
* Patient or patient's representative provides consent
* Pre-stroke modified Rankin Scale (mRS) of < =2
* General endotracheal anesthesia (GETA) is planned to be used, as standard care, for IAMT
* Treatment with iNO requires mechanical ventilation. Because IAMT can be performed using conscious sedation and not GETA, only those patients for which the procedure is planned with GETA will be included. The decision for the type of anesthetic depends on the severity of stroke, region of brain affected by the stroke, and the ability for the patient to cooperate for the procedure.

Exclusion Criteria:

* Hypotension at presentation, defined as systolic blood pressure (SBP) < 100 or MAP < 60; profound hypertension with SBP >185 or DBP >110mmHg unable to be controlled with IV medications
* Inability to undergo a brain MRI (e.g., implanted pacemaker)
* Patients who received IV tPA >4.5hrs after symptom onset
* Coaguloapathy, defined as platelet count < 50,000, INR >3.0, PTT > 3x normal, use of novel anticoagulants with eGFR < 30ml/min
* Vulnerable Subjects including: mentally ill or incompetent patients, those with diminished decision-making capacity, prisoners, inpatient care for long-term chronic illness, terminally ill, pregnant women, and children
* Any form of hemorrhage on non-contrast CT Head or mass lesion
* Severe head injury within 90 days
* Pre-existing severe neurological/psychiatric disease
* Seizure at stroke onset (unable to assess NIHSS)
* Blood glucose < 50mg/dL or >400mg/dL
* Hemoglobin <7mmol/L
* eGFR < 30ml/min
* Allergy to contrast media
* Presumed septic embolus as source of stroke
* Flow limiting intracranial or extracranial carotid stenosis, or complete carotid occlusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Maximum safe dose of iNO for AIS patients - assessing for reperfusion hemorrhage/symptomatic intracranial hemorrhage (sICH) | Year 2
  To establish a maximum safe dose of iNO for acute ischemic (non-bleeding) stroke (AIS) patients, assessing for reperfusion hemorrhage/symptomatic intracranial hemorrhage (sICH)

SECONDARY OUTCOMES:
Change in pre-endovascular mechanical thrombectomy (IAMT) and post-IAMT core infarct volume | Year 2
  Core infarct measurement pre/post

CONTACTS AND LOCATIONS:
Overall Officials: William R Stetler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Carolinas Medical Center, Charlotte, North Carolina
  - Atrium Health, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No